CLINICAL TRIAL: NCT03351686
Title: The Effect of Tranexamic Acid in Preventing Postpartum Hemorrhage in High Risk Pregnancies During Elective Cesarean Section, a Randomized Controlled Clinical Trial
Brief Title: Tranexamic Acid in Preventing Postpartum Hemorrhage in High Risk Pregnancies During Elective Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hanan Nabil, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MansuraU
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Postpartum Hemorrhage
Keywords: tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid group (Experimental)
  Interventions: Drug: Tranexamic Acid
- non tranexamic (control) group (No Intervention)

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid (Kepron, Amoun, Egypt) was given slowly intravenously over 10 minutes just before the skin incision of elective cesarean section to group A. Tranexamic acid injection was prepared by diluting 1g (10 mL) tranexamic acid into 20 ml of 5% glucose.
  Arms: tranexamic acid group

SUMMARY:
postpartum hemorrhage (PPT) represents one of the major causes of maternal mortality . Tranexamic acid is used in many studies in management of PPH in combination with ecobolics. this study aims to evaluate the possible value of the use of tranexamic acid in prevention of postpartum hemorrhage .

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 28 weeks or more.
* Chronic Hypertension.
* Preeclapmsia -Eclampsia.
* Multiple pregnancy.
* Uterine Liomyomas.
* Polyhydraminos.
* Fetal macrosomia.
* Associated Thrombocytopenia
* History of postpartum hemorrhage.

Exclusion Criteria:

* Patients with rheumatic heart disease.
* Patients with history Cardiac Valve Replacement.
* Current or past history of DVT.
* Women on any anticoagulant therapy.
* Sensitivity to tranexamic acid
* Pregnancies with any abnormally implanted or located placenta.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
prevention of postpartum hemorrhage in high risk group | intraoperative
  assessment of intraoperative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Nabil, MD, Principal Investigator — Mansoura University